CLINICAL TRIAL: NCT02779153
Title: Efficacy, Safety, and Steroid Sparing Effect of Acthar in Patients With Hematologic Manifestations of Systemic Lupus Erythematosus
Brief Title: Acthar SLE (Systemic Lupus Erythematosus)
Acronym: Acthar SLE
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: closed in agreement of the sponsor and institution due to lack of patient accrual.
Sponsor: NYU Langone Health (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-00295
Record Dates: First submitted 2016-05-18; First posted 2016-05-20 (Estimated); Last update posted 2019-09-13 (Actual); Status verified 2019-09

CONDITIONS: Systemic Lupus Erythematosus (SLE); Repository Corticotropin Injection
Keywords: SLE; H.P. Acthar Gel
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Adrenocorticotropic Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acthar low dose (40 U) (Experimental)
  Interventions: Drug: Acthar low dose (40 U)
- Acthar high dose (80 U) (Experimental)
  Interventions: Drug: Acthar high dose (80 U)

INTERVENTIONS:
Drug: Acthar low dose (40 U) — The 40U group will administer 0.5 mL of study medication once a day. Patients will taper study medication during Week 2 through the remainder of the study and will administer 0.5 mL of study medication twice a week. The stable Acthar regimen should be maintained for the remainder of the study. However, dose adjustments may be implemented if needed based on safety.
  Other Names: Repository Corticotropin Injection
  Arms: Acthar low dose (40 U)
Drug: Acthar high dose (80 U) — The 80U group will administer 1.0 mL of study medication every day. If a patient meets dose reduction criteria, their assigned volume will be adjusted from 1.0 mL to 0.5 mL. Patients will taper study medication during Week 2 through the remainder of the study. However, dose adjustments may be implemented if needed based on safety.
  Other Names: Repository Corticotropin Injection
  Arms: Acthar high dose (80 U)

SUMMARY:
This is a randomized study exploring the efficacy, safety and steroid sparing ability of two doses (40 U and 80 U) of Acthar in SLE patients with immune mediated hematologic manifestations requiring steroid use for a minimum of 2 weeks prior to screening.

DETAILED DESCRIPTION:
Acthar is currently labeled for use during an exacerbation or for maintenance therapy in selected SLE cases, however data from prospective trials on hematologic manifestations of SLE are not available. Due to the potential effect of lowering or eliminating autoantibodies, the absence of bone marrow suppression, and a steroid sparing effect, Acthar may represent a novel therapeutic option in recalcitrant cases of hematologic SLE.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent.
* Diagnosis of SLE according to the American College of Rheumatology revised criteria (fulfilled ≥ 4 criteria).
* Hematologic BILAG scores due to hemolytic anemia or thrombocytopenia of BILAG A (including hemolytic anemia with hemoglobin < 8.0 g/dL or platelet count < 25 x 109 l) or BILAG B (including hemolytic anemia with hemoglobin 8.0 - 9.9 g/dDL or platelet count 25 - 49 x 109 l) based on screening laboratory assessment.
* Currently taking prednisone ≥ 7.5 mg or equivalent for hematologic SLE for at least 2 weeks prior to screening.
* Use of antimalarials and NSAIDs (stable regimen within the 4 weeks prior to screening), as well as methotrexate, azathioprine, and mycophenolate mofetil (stable regimen within the 4 weeks prior to screening) are permitted but not required. If used, the regimen must remain stable through the study. An increase or addition of SLE medication at any time during the study is not permitted.
* Ability to comply with study procedures, which include SC injections of study medication, adhering to concomitant medication restrictions, and attending scheduled office visits.

Exclusion Criteria:

* Patients with a recent history (< 2 week prior to screening) of starting prednisone or equivalent.
* Patients with active nephritis, defined as serum creatinine > 2.5 mg/dL or protein/creatinine ratio (PCR) > 1.5 g/g, or patients that required hemodialysis within 3 months prior to screening.
* Active central nervous system (CNS) lupus (including seizures, psychosis, organic brain syndrome, cerebrovascular accident, cerebritis, or CNS vasculitis), requiring therapeutic intervention within 3 months prior to screening.
* Type 1 or type 2 diabetes mellitus (history of gestational diabetes is not an exclusion), or patients currently taking hypoglycemic medication.
* Patients with a history of concomitant medication use as follows:

  a. Receipt of the following within 1 month prior to screening: i. Any steroid injection (IM, intraarticular, or IV) b. Receipt of any of the following within 3 months prior to screening: i. Cyclosporine ii. Any non-biologic investigational drug c. Receipt of the following within 4 months prior to screening: i. IVIg ii. Plasmapheresis d. Receipt of cyclophosphamide within 6 months prior to screening e. Receipt of the following within 12 months prior to screening: i. B cell targeted therapy (rituximab or other anti-CD20 agent, anti-CD22 [epratuzumab], anti-CD52 [alentuzumab], or belimumab) ii. Abatacept iii. Any biologic investigational agent
* Contraindication per Acthar Prescribing Information: scleroderma, osteoporosis, systemic fungal infections, ocular herpes simplex, recent surgery, history of or the presence of peptic ulcer, congestive heart failure, uncontrolled hypertension, primary adrenocortical insufficiency, or adrenal cortical hyperfunction.

  1. For the purposes of this study, osteoporosis is defined as evidence of vertebral or long bone fracture, or lumbar spine T-score > 2.0 standard deviations below the mean of the reference population.
  2. For the purposes of this study, history of peptic ulcer is defined as ≤ 6 months prior to screening.
  3. For the purposes of this study, congestive heart failure is defined as New York Heart Association Functional Class III-IV.
  4. For the purposes of this study, uncontrolled hypertension is defined as a mean systolic blood pressure ≥ 140 mm Hg and/or diastolic blood pressure ≥ 90 mm Hg on ≥ 3 seated readings taken at least 5 minutes apart during the screening period.
* Reproductive status:

  1. Women who are pregnant,
  2. Women who are breastfeeding,
  3. Women of childbearing potential who are unwilling or unable to use an acceptable method of birth control to avoid pregnancy for the entire study period, as evaluated by the Investigator (women of non-childbearing potential are those that have a history of hysterectomy, bilateral oophorectomy, or are postmenopausal with no history of menstrual flow for ≥ 12 months prior to screening).
* Immune System: Known immunocompromised status (not related to SLE or therapies for SLE), including individuals who have undergone organ transplantation or who are known to be positive for the human immunodeficiency virus.
* Patients with acute or chronic hepatitis C, or active hepatitis B infection, positive interferon gamma release assay (IGRA) or signs or symptoms concerning for active tuberculosis (TB); or use of antibiotics (antibacterial, antiviral, antifungal, or antiparasitic agent) within 4 weeks of randomization for treatment of an active infection.
* Presence of any other clinically significant disease or disorder which, in the opinion of the Investigator (by its nature or by being inadequately controlled), might put the patient at risk due to participation in the study, or may influence the results of the study or the patient's ability to complete the study.
* Any clinically significant laboratory abnormality, based on the Investigator's judgment. The following laboratory exclusions apply for all patients:

  1. AST > 2.5 times the upper limit of normal (ULN)
  2. ALT > 2.5 times ULN
  3. Hemoglobin A1c > 6.5%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-10; Primary Completion 2019-05-22 (Actual); Study Completion 2019-05-22 (Actual)

PRIMARY OUTCOMES:
Systemic Lupus Erythematosus Disease Activity Index (SLEDAI) Score | Baseline to Week 24
  Disease activity is based on 24 questions, weighted across nine organ systems, combined into a total score that can range from 0 to 105, but are generally < 20, even with very active disease.
British Isles Lupus Assessment Group (BILAG) disease activity index Score | Baseline to Week 24
  Items are rated as 0 (not present), 1 (improving), 2 (same), 3 (worse), or 4 (new) in the last 4 weeks compared with the previous 4 weeks. The numerical scores are used to categorize each organ system by an alphabetical score: 'A' reflecting severe disease requiring increases in prednisone to > 20 mg daily and/or addition of immunosuppressive agents, 'B' indicated less active disease, requiring low-dose prednisone and/or symptomatic treatment with NSAIDs and/or antimalarials, 'C' reflecting mild disease requiring only symptomatic therapy, 'D' reflecting previous organ system involvement without current disease activity, and 'E' reflecting no prior or no current disease involvement in that organ system.
Physician's Global Assessment Score | Baseline to Week 24
  The Physician's Global Assessment is a 10 cm visual analogue scale (VAS) anchored at 0 (none) and 3 (severe) with intermediate lines at 1 (mild) and 2 (moderate). It is designed for the physician to indicate the patient's overall disease activity at a particular visit
SELENA Flare Index Score | Baseline to Week 24
  The SELENA Flare Index categorizes SLE flare as 'mild or moderate' or 'severe' based on six variables
  * Change in SLEDAI score from the most recent assessment to current.
  * Change in signs or symptoms of disease activity.
  * Change in prednisone dosage.
  * Use of new medication for disease activity or hospitalization.
  * Change in PGA score.
  * Hospitalization for SLE activity (severe flare only).
SLICC/ACR Damage Index | Baseline to Week 24
  The SLICC/ACR Damage Index measures irreversible organ damage from either the disease process or treatment, which has been present for ≥ 6 months, in 12 organ systems. It is an important predictor of long-term mortality and is an independent outcome measure separate from the SLEDAI.

SECONDARY OUTCOMES:
Medical Outcomes Survey Short Form-36 | Baseline to Week 24
  The SF-36 has been validated in SLE and includes eight domains: physical functioning, role physical, bodily pain, general health perceptions, vitality (which includes fatigue, energy and vigor), social functioning, role emotional and mental-health impact, combined into two summary scores (physical component summary scores [PCS] and mental component summary scores [MCS])
FACIT Fatigue Scale | Baseline to Week 24
  The FACIT-F scale is a 13-item questionnaire to evaluate self-reported fatigue and its impact upon daily activities and function. The responses are measured on a 4-point Likert scale, with the total score ranging from 0 to 52. The FACIT-F scale has been validated in SLE patients.
Patient's Global Assessment | Baseline to Week 24
  Subjects rate their global assessment of SLE disease activity on each visit, in response to the question "Considering all the ways your SLE affects you, please mark a vertical line on the scale below for how are you feeling today?" using a 100mm visual analogue scale, where 0 is "very good, no symptoms" and 100 is "very poor, very severe symptoms."

CONTACTS AND LOCATIONS:
Overall Officials: Amit Saxena, MD, Principal Investigator — New York University Medical School